CLINICAL TRIAL: NCT06857058
Title: A Prospective, Multicenter, Registry Study to Evaluate the Safety, Efficacy, and Standardized Procedural Optimization of the Intracranial Drug-Eluting Stent System in Patients with Symptomatic Intracranial Atherosclerotic Stenosis
Brief Title: Standardized Procedure for Intracranial Drug-Eluting Stenting in the Treatment of Intracranial Atherosclerotic Stenosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sino Medical Sciences Technology Inc. (Industry)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); Tongji Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SN-NOVA II SOP-202501
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-02

CONDITIONS: Intracranial Atherosclerotic Stenosis
Keywords: endovascular therapy, intracranial drug-eluting stent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NOVA DES (Experimental): Patients who met the inclusion criteria were implanted with the NOVA stent, and the procedure was documented in detail.
  Interventions: Device: NOVA DES

INTERVENTIONS:
Device: NOVA DES — The NOVA stent is a sirolimus-eluting stent system designed for intracranial artery stenosis with a rapid exchangeable balloon

SUMMARY:
The primary objective of this trial is to evaluate the Safety, Efficacy, and Standardized Procedural Optimization of the Intracranial Drug-Eluting Stent System in Patients with Symptomatic Intracranial Atherosclerotic Stenosis.

DETAILED DESCRIPTION:
The investigation is a prospective, multi-center clinical study. The trial is expected to enroll 300 subjects. The population for this study is subjects with intracranial atherosclerotic stenosis who are suitable candidates for stent angioplasty. Patients fulfilling all of the inclusion criteria and none of the exclusion criteria will be enrolled after they signed the informed consent form. The study consists of ten visits including preoperative screening, procedure date, 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years. The primary endpoints are stroke or death within 30 days after enrollment, plus any ischemic stroke or revascularization from the original culprit intracranial artery beyond 30 days through 12 months after procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between 18 and 80 years of age
2. Symptomatic intracranial arteriosclerosis stenosis with reference diameter 2.25-4.00mm
3. Intracranial artery stenosis ( ≥70%) conformed by DSA
4. Those who voluntarily participate in the study and sign informed consent form

Exclusion Criteria:

1. Those who have surgery within previous 30 days or plan to perform major surgery in the next 90 days (surgery grade 3 and above);
2. Subjects of acute hemorrhagic stroke within 3 months;
3. The baseline mRS of disabling stroke is more than 3;
4. The target vessel is severely calcified and closely related to stenosis;
5. Non-atherosclerotic diseases (e.g. arterial dissection, Moya Moya disease, vascular inflammatory lesions caused by infection, autoimmune diseases, post-irradiation, postpartum status; developmental or genetic abnormalities such as fibromuscular dysplasia, sickle cell anemia, suspected vasospasm);
6. It is suspected that the ischemic event is due to embolism or arterial embolism from the extracranial segment (including ipsilateral chest or neck vascular occlusive disease) or potential cardiogenic embolism (e.g. atrial fibrillation, mitral stenosis, patent foramen ovale, left ventricular thrombus, myocardial infarction within 6 weeks, etc.);
7. The presence of a >50% stenosis in the main blood supply artery of the target vessel. For example, when the lesion is located in the middle cerebral artery, the ipsilateral internal carotid artery stenosis by over 50% should be excluded; when the lesion is located in the basilar artery, the dominant side vertebral artery stenosis >50% should be excluded;
8. There are intracranial tumors, or intracranial arteriovenous malformations;
9. Those who are allergic to heparin, aspirin, clopidogrel, contrast agents, anesthetics, and stent components;
10. Pregnant and lactating women
11. Those who are unable to complete follow-up because of mental illness, cognitive or emotional disorders;
12. Inapplicable for this study at the investigators' viewpoints.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2026-06-08 (Estimated); Study Completion 2026-06-08 (Estimated)

PRIMARY OUTCOMES:
Stroke or death within 30 days after enrollment, plus any ischemic stroke or revascularization from the original culprit intracranial artery beyond 30 days through 12 months after procedure. | 1 year after procedure
  This outcome includes ischemic/hemorrhagic stroke and all-cause death within 30 days after procedure of the qualifying lesion during follow-up, or any ischemic stroke and revascularization from the original culprit symptomatic intracranial artery beyond 30 days through 12 months after procedure.

SECONDARY OUTCOMES:
Rate of any stroke (hemorrhagic/ischemic stroke) in the target blood supply area or all-cause death at 30 days after procedure | 30 days after procedure
  The rate of Hemorrhagic stroke as well as symptomatic ischemic stroke and any death in the target blood supply area
Rate of any stroke (hemorrhagic/ischemic stroke) in the non-target blood supply area or all-cause death at 30 days after procedure | 30 days after procedure
  The rate of Hemorrhagic stroke as well as symptomatic ischemic stroke and any death in the non-target blood supply area
Rate of TIA at 30 days, 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after procedure | 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after procedure
  TIA is a temporary blockage of blood flow to the brain with symptoms last from only a few minutes up to 24 hours
Rate of any stroke (hemorrhagic/ischemic stroke) in the target blood supply area at 3, 6 months, 1, 2, 3, 4 years and 5 years after procedure | 3, 6 months, 1, 2, 3, 4 years and 5 years after procedure
  The rate of Hemorrhagic stroke as well as symptomatic ischemic stroke in the target blood supply area
Rate of any stroke (hemorrhagic/ischemic stroke) in the non-target blood supply area at 3, 6 months, 1, 2, 3, 4 years and 5 years after procedure | 3, 6 months, 1, 2, 3, 4 years and 5 years after procedure
  The rate of Hemorrhagic stroke as well as symptomatic ischemic stroke in the non-target blood supply area
Rate of death (vascular/ non-vascular death) at 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after procedure | 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after procedure
  The cause of death was classified as vascular or nonvascular and based on information obtained from the family, medical records, and death certificates. Vascular death included death due to stroke, MI, heart failure, pulmonary embolus, cardiac arrhythmia, or other vascular cause.
Rate of symptomatic ISR and Revascularization at 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after procedure | 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after procedure
  symptomatic ISR is defined as ISR associated with an ischemic event in the territory. Revascularization is the restoration or improvement of blood supply, and included surgical operation, endovascular procedures, etc.
Rate of modified Rankin Scale (mRS) at 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after procedure | 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after procedure
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6 with "0" being perfect health without symptoms to "6" being death.
EQ-5D score at 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after procedure | 30 days, 3, 6 months, 1, 2, 3, 4 years and 5 years after procedure
  A health state defined by the descriptive EQ-5D system can be described by a five-digit number, each digit indicating the score of the corresponding dimension.
Rate of in-stent restenosis at 1, 2, 3, 4 years and 5 years after procedure (Optional) | 1, 2, 3, 4 years and 5 years after procedure
  Patients with ≥50% stenosis of the vessel
Rate of Device defect | within 5 years of whole trial
  Device defects refer to the unreasonable risks that may endanger human health and life safety during the normal use of medical devices in the course of clinical trials, such as label errors, quality problems, failures, etc.
Rate of bleeding events at 1 years after procedure | 1 year after procedure
  Bleeding was defined according to Bleeding Academic Research Consortium

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Guan, Principal Investigator — The First Affiliated Hospital of Zhengzhou University; Chun Fang, Principal Investigator — Tongji Hospital
Locations (1):
- The first affiliated hospital of zhengzhou university, Zhengzhou, China